CLINICAL TRIAL: NCT04741503
Title: Project Insight: Feasibility of a Breast Cancer Screening Decision Support Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202101073; 5R00MD011485-04 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-02-05 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer Screening; Oncology; Preventative Medicine; Mammography
Keywords: Health Literacy; Health Disparities; Shared Decision Making
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast Cancer Screening Decision Support Tool (Experimental): -After randomization, participants will complete pre-questionnaires, review the Breast Cancer Screening Decision support tool, and then complete the post-questionnaire.
  Interventions: Other: Breast Cancer Screening Decision Support Tool
- Standard Breast Cancer Screening Education (Active Comparator): -After randomization, participants will complete pre-questionnaires, review the standard breast cancer screening education from the NCI, and then complete the post-questionnaire.
  Interventions: Other: National Cancer Institute Breast Cancer Screening PDQ

INTERVENTIONS:
Other: Breast Cancer Screening Decision Support Tool — -Provides a description of screening mammography, current screening recommendations, benefits and downsides, narratives, and questions for the participant's physician.
  Arms: Breast Cancer Screening Decision Support Tool
Other: National Cancer Institute Breast Cancer Screening PDQ — -Provides current information about breast cancer screening and is meant to inform and help patients
  Arms: Standard Breast Cancer Screening Education

SUMMARY:
The purpose of this investigation is to conduct a feasibility study to evaluate the potential for implementing the developed decision support tool with Latina, Black, and non-Latina White women. The investigators will collect feasibility data and assess the use of the decision support tool with end-users. The aim is to determine if women using the decision support tool make more informed choices measured by knowledge, attitudes, and intentions.

ELIGIBILITY:
Inclusion Criteria:

* Latina, Black, or non-Latina White women
* Between the ages of 40-49 years
* Can write, read, and understand English

Exclusion Criteria:

-Women with greater than an average self-reported risk of breast cancer will be ineligible for participation, as evidenced by any of the following:

* Self-reported personal history of breast cancer (invasive, ductal carcinoma in situ [DCIS], or lobular carcinoma in situ[LCIS])
* Self-reported personal history of atypical hyperplasia
* Self-reported first degree family member with history of breast cancer (e.g., mother, sister)
* Self-reported known underlying genetic mutation such as a BRCA1/BRCA2 gene
* Self-reported prior thoracic or chest wall radiation therapy

Ages: 40 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1277 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley J Housten, OTD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after De-identified data may be shared upon reasonable request.
Time Frame: Up to 36 months following publication
Access Criteria: Please contact the principal investigator with requests.

REFERENCES:
- [Derived] Riganti P, Ruiz Yanzi MV, Escobar Liquitay CM, Sgarbossa NJ, Alarcon-Ruiz CA, Kopitowski KS, Franco JV. Shared decision-making for supporting women's decisions about breast cancer screening. Cochrane Database Syst Rev. 2024 May 10;5(5):CD013822. doi: 10.1002/14651858.CD013822.pub2. PMID 38726892
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1277 participants consented to participate in the study. 767 participants were removed prior to randomization as they failed to meet screening criteria. 186 participants were removed prior to randomization as overquotas (i.e., having already met the targeted goals for race/ethnicity) were removed.
Groups:
- Participants Who Were Not Randomized: Participants who consented to participate in the study but were removed prior to randomization.
Period: Initial Enrollment
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education | Participants Who Were Not Randomized
Started | 160 | 164 | 953
Completed | 160 | 164 | 0
Not Completed | 0 | 0 | 953
Not completed — Failed to meet screening criteria | 0 | 0 | 767
Not completed — Overquotas removed | 0 | 0 | 186
Period: Met Protocol Criteria for Data Inclusion
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education | Participants Who Were Not Randomized
Started | 160 | 164 | 0
Completed | 137 | 147 | 0
Not Completed | 23 | 17 | 0
Not completed — Removed from study for not meeting protocol criteria for free responses to knowledge questions | 23 | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education | Total
Number analyzed (Participants) | 160 | 164 | 324
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 160 | 164 | 324
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 164 | 324
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 52 | 98
  Not Hispanic or Latino | 114 | 111 | 225
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 61 | 112
  White | 81 | 72 | 153
  More than one race | 13 | 12 | 25
  Unknown or Not Reported | 10 | 17 | 27
Region of Enrollment [Number; unit: participants]
  United States | 160 | 164 | 324

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Knowledge Score of Screening Mammography Guidelines
Description: * The total knowledge score will be collected by the Breast Cancer and Breast Cancer Screening Mammography knowledge questions.
  * This questionnaire was modified from an existing breast cancer screening knowledge from Hersch et al. This questionnaire covers mammography, screening benefits and downsides, and guidelines.
  * Six of the knowledge questions were scored as correct (1) or incorrect/unsure (0). The percentage of correct scores was calculated per participant pre-intervention and post-intervention (range, 0-100). A higher score indicates higher knowledge.
Time Frame: In both the pre-questionnaire and post-questionnaires occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
score on a scale
  Pre-questionnaire | 51.0 (26.1) | 47.0 (26.4)
  Post-questionnaire | 56.2 (28.6) | 54.6 (29.3)

2. Primary Outcome: Feelings of Being Fully Informed and Clear About the Importance of the Components for Making Informed Decisions as Measured by the Decisional Conflict Scale (DCS), Values Clarity Subscale
Description: -The 3-item Values Clarity Subscale (questions 4-6) uses a 5-point response format, ranging from 0 (yes) to 4 (no) to assess feelings of clarity about personal values for benefits and risks/side effects. Items are summed and scores are calculated on a range of 0 (feels extremely clear about personal values for benefits/risks) to 100 (feels extremely unclear about personal values). A higher score indicates less clarity on personal values.
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
score on a scale | 19.6 (19.7) | 16.4 (19.5)

3. Primary Outcome: Decision Self-efficacy as Measured by the 5-Point Decision Self-Efficacy Scale
Description: -The 5-Point Decision Self-Efficacy Scale will be modified for breast cancer screening and will measure self-confidence or belief in one's decision-making abilities, including shared decision-making. Questions ask participants how confident they are in a variety of health related skills. This 11-item scale has five response options from "not at all confident" (0) to "extremely confident" (4). Items are summed and scores are calculated on a range of 0-100. A higher score indicates higher decisional self-efficacy.
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
score on a scale | 69.2 (20.2) | 73.2 (21.1)

4. Primary Outcome: Preparation for Decision Making Scale as Measured by PrepDM
Description: -The Preparation for Decision Making Scale (PrepDM) assesses a patient's perception of how useful a decision aid or educational materials are in making a screening or treatment decision. The 10-item scale uses a 5-point Likert response format, ranging from 0 (not at all) to 4 (a great deal). Items are summed and scores are calculated on a range of 0-100. Higher scores indicate higher perceived levels of preparation for decision making.
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
score on a scale | 69.2 (21.9) | 68.5 (27.0)

5. Secondary Outcome: Acceptability as Measured by the Ottawa Acceptability Measures - Presented Information
Description: -Adapted acceptability measures from the Ottawa Acceptability Measures including questions eliciting ratings of the information presented in the tool. Each question will ask the participant to rate the information in the tool they viewed as poor, fair, good, or excellent to show what they thought about the way the information was presented.
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Population: Stories about other women question was only asked of the Breast Cancer Screening Decision Support Tool arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
Participants
  Breast cancer: Poor | 2 | 7
  Breast cancer: Fair | 29 | 19
  Breast cancer: Good | 66 | 73
  Breast cancer: Excellent | 40 | 47
  Breast cancer: Missing responses | 0 | 1
  Breast cancer screening mammography: Poor | 2 | 7
  Breast cancer screening mammography: Fair | 22 | 15
  Breast cancer screening mammography: Good | 66 | 72
  Breast cancer screening mammography: Excellent | 47 | 53
  Breast cancer screening mammography: Missing responses | 0 | 0
  Guidelines for screening: Poor | 1 | 5
  Guidelines for screening: Fair | 23 | 17
  Guidelines for screening: Good | 63 | 78
  Guidelines for screening: Excellent | 50 | 47
  Guidelines for screening: Missing responses | 0 | 0
  Benefits of screening: Poor | 1 | 4
  Benefits of screening: Fair | 20 | 15
  Benefits of screening: Good | 63 | 66
  Benefits of screening: Excellent | 53 | 62
  Benefits of screening: Missing responses | 0 | 0
  Downsides of screening: Poor | 4 | 8
  Downsides of screening: Fair | 30 | 34
  Downsides of screening: Good | 61 | 64
  Downsides of screening: Excellent | 42 | 41
  Downsides of screening: Missing responses | 0 | 0
  Questions to help make the decision: Poor | 2 | 4
  Questions to help make the decision: Fair | 26 | 20
  Questions to help make the decision: Good | 63 | 77
  Questions to help make the decision: Excellent | 46 | 46
  Questions to help make the decision: Missing responses | 0 | 0
  Stories about other women: number analyzed (Participants) | 137 | 0
  Stories about other women: Poor | 2 |
  Stories about other women: Fair | 29 |
  Stories about other women: Good | 67 |
  Stories about other women: Excellent | 39 |
  Stories about other women: Missing responses | 0 |

6. Secondary Outcome: Acceptability as Measured by the Ottawa Acceptability Measures - Length of Tool
Description: -Adapted acceptability measures from the Ottawa Acceptability Measures eliciting acceptability ratings of the length of tool. The questionnaire asks the participant to rate the length of the tool they viewed as too long, too short, just right, or prefer not to answer.
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
Participants
  Too long | 16 | 33
  Too short | 4 | 6
  Just right | 113 | 105
  Prefer not to answer | 4 | 3

7. Secondary Outcome: Acceptability as Measured by the Ottawa Acceptability Measures - Amount of Information
Description: -Adapted acceptability measures from the Ottawa Acceptability Measures eliciting acceptability ratings of the amount of information in the tool. The questionnaire asks the participant to rate the amount of information as too much information, too little information, just right, or prefer not to answer.
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
Participants
  Too much information | 11 | 19
  Too little information | 18 | 15
  Just right | 105 | 109
  Prefer not to answer | 3 | 4

8. Secondary Outcome: Acceptability as Measured by the Ottawa Acceptability Measures - Tool's Balance
Description: -Adapted acceptability measures from the Ottawa Acceptability Measures eliciting acceptability ratings of the balance of the tool's balance. The questionnaire asks the participant to rate the tool as slanted towards screening, slanted towards NOT screening, balanced, or prefer not to answer
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
Participants
  Slanted towards screening | 30 | 31
  Slanted towards NOT screening | 4 | 5
  Balanced | 98 | 103
  Prefer not to answer | 3 | 8

9. Secondary Outcome: Acceptability as Measured by the Ottawa Acceptability Measures - Usefulness of Tool
Description: -Adapted acceptability measures from the Ottawa Acceptability Measures eliciting acceptability ratings of the usefulness of the tool for decision-making. The questionnaire asks the participant if they would find this decision tool useful when making decision for when to start screening mammography (yes, no, prefer not to answer).
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
Participants
  Yes | 114 | 119
  No | 17 | 20
  Prefer not to answer | 6 | 8

10. Secondary Outcome: Acceptability as Measured by the Ottawa Acceptability Measures - Helpfulness of Tool for Decision Making
Description: -Adapted acceptability measures from the Ottawa Acceptability Measures eliciting acceptability ratings of the helpfulness for decision making of the breast cancer screening decision support tool's questions. The questionnaire asks the participant if the questions in the tool made decision making easier or more difficult or if they prefer not to answer.
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Population: This question was for participants enrolled in the Breast Cancer Screening Decision Support Tool arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 0
Participants
  Easy | 119 |
  Difficult | 7 |
  Prefer not to answer | 10 |

11. Secondary Outcome: Acceptability as Measured by the Ottawa Acceptability Measures - Amount of Information for Decision Making
Description: -Adapted acceptability measures from the Ottawa Acceptability Measures eliciting acceptability ratings of the amount of information in the tool for decision making. The questionnaire asks the participant if the tool provided enough information to help a woman decide when to start breast cancer screening mammography (yes, no, prefer not to answer).
Time Frame: In the post-questionnaire occurring in a single encounter in one day (Day 1 approximately 30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
Participants
  Yes | 125 | 129
  No | 10 | 13
  Prefer not to answer | 2 | 5

12. Secondary Outcome: Intention to Screen
Description: -This is the participants' intention to undergo breast cancer screening within the upcoming year. The questionnaire asks the participant how likely they are to have a screening mammography this upcoming year. Response options include: leaning toward screening (definitely will be tested or probably will be tested), leaning away from screening (probably won't be tested or definitely won't be tested), unsure, and prefer not to answer.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
Number analyzed (Participants) | 137 | 147
Participants
  Pre-questionnaire: Leaning toward screening | 95 | 104
  Pre-questionnaire: Leaning away from screening | 17 | 24
  Pre-questionnaire: Unsure or unknown (no response) | 25 | 19
  Post-questionnaire: Leaning toward screening | 96 | 103
  Post-questionnaire: Leaning away from screening | 16 | 27
  Post-questionnaire: Unsure or unknown (no response) | 25 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were followed through completion of questionnaires (day 1 - approximately 30 minutes)
Arm/Group | Breast Cancer Screening Decision Support Tool | Standard Breast Cancer Screening Education
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/147
Other Adverse Events (participants affected / at risk) | 0/137 | 0/147

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04741503/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT04741503/ICF_001.pdf